CLINICAL TRIAL: NCT02939508
Title: Acute Lower Gastrointestinal Dysfunction in Critical Care Patients: Should Colon or Non-colon Originated Lesions be Distinguished?
Brief Title: Should Colon or Non-colon Originated Lesions be Distinguished?
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Medical Association (Network)
Responsible Party: Principal Investigator, Juanhong Shen, Director, PhD, Principal Investigator, Resident Physician, Chinese Medical Association
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Jinling37ICUZCY
Record Dates: First submitted 2016-10-07; First posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Acute Lower Gastrointestinal Dysfunction
Keywords: Acute lower gastrointestinal dysfunction; Colon-originated lesions; Critical patient; Colonoscopic decompression; Anticholinergic drugs
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colon originated (Experimental): A history of colon (-innervating) nerve damage, moderate or more severe edema; and without a history of colon (-innervating) nerve damage, with mild or severe edema of colonic wall on CT.
  Interventions: Other: Colon originated: Neostigmin, Colonoscopy decompression, Surgery
- Non-colon originated (Active Comparator): NCOG met one of the two following criteria:
  1. History of nerve damage that could affect colon movement (colon [-innervating] nerve damage), such as pelvic or retroperitoneal operation, spine injury, or cerebral lesion; and non-existing or mild edema of colonic wall on abdominal CT;
  2. Absence of history of colon(-innervating) nerve damage, with no obvious change in the colonic wall visible on the CT scan.
  Interventions: Other: Non-colon originated: Neostigmin, Colonoscopy decompression

INTERVENTIONS:
Other: Colon originated: Neostigmin, Colonoscopy decompression, Surgery
  Arms: Colon originated
Other: Non-colon originated: Neostigmin, Colonoscopy decompression
  Arms: Non-colon originated

SUMMARY:
This prospective study was designed to compare the difference of effects of conventional treatment, medicine intervention, endoscopic therapy, and surgery between colon originated and non-colon originated ALGID in critical patients, in order to alert doctors to differ the treatment of the two ALGID and provide basis for treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in our ICU aged 18-75 years.
2. Patients with a confirmed diagnosis of ALGID.

Exclusion Criteria:

1. mechanical intestinal obstruction (including tumor, stercoral obstruction etc.)
2. gastrointestinal hemorrhage within 72 hours.
3. history of inflammatory bowel disease (ulcerative colitis or Crohn's disease) or radiation enteritis.
4. pregnancy.
5. contraindications of neostigmine administration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
28-day mortality after admission | 1-28 day after admission
ICU mortality, n (%) | 1-28 day after ICU admission

SECONDARY OUTCOMES:
ICU stage, (day) | 1-60 day after ICU admission
Hospitalization, (day) | 1-60 day after admission
intra-abdominal pressure | 1-28 day after admission
Abdominal compartment syndrome | 1-28 day after admission

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided